CLINICAL TRIAL: NCT01601366
Title: Levonorgestrel-releasing Intrauterine System Compared to Low Dose Combined Oral Contraceptive Pills for Treatment of Adenomyosis: a Randomized Controlled Trial
Brief Title: LNG-IUS for Treatment of Dysmenorrhea
Acronym: LNGIUSAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omar Mamdouh Shaaban (Other)
Responsible Party: Sponsor-Investigator, Omar Mamdouh Shaaban, Dr., Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNG-IUS-dysmenorrhea; AUM001206
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; Intrauterine levonorgestrel; Dysmenorrhea; Oral contraceptives; Uterus
MeSH Terms: conditions — Adenomyosis; Dysmenorrhea | interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LNG-IUS (Mirena) (Experimental): Group I "the LNG-IUS group" where they will have a LNG IUS (mirena) inserted for them
  Interventions: Device: LNG-IUS
- Combined oral contraceptives (Active Comparator): Group II "COCs group" where they will receive low dose combined oral contraceptive pills for 6 months
  Interventions: Drug: Combined oral contraceptives

INTERVENTIONS:
Device: LNG-IUS — The study includes 2 treatment groups: Group I "the LNG-IUS group" where they will have a LNG IUS inserted for them
  Other Names: Mirena
  Arms: LNG-IUS (Mirena)
Drug: Combined oral contraceptives — Group II: will recite combined oral contraceptives for 6 months
  Other Names: Gynera
  Arms: Combined oral contraceptives

SUMMARY:
Adenomyosis is a disease entity diagnosed when endometrial glands and stroma deep in the myometrium are associated with surrounding myometrial hypertrophy. The finding classically associated with adenomyosis is excessive uterine bleeding accompanied by worsening dysmenorrhea. The advent of endovaginal US has substantially improved the ability to diagnose adenomyosis. Different US features of adenomyosis have been reported, including uterine enlargement not explainable by the presence of leiomyomas, asymmetric thickening of the anterior or posterior myometrial wall, lack of contour abnormality or mass effect, heterogeneous poorly circumscribed areas within the myometrium, anechoic lacunae or cysts of varying sizes, and increased echotexture of the myometrium.

Transvaginal power Doppler application is useful in studying the vascular tree of adenomyosis and can aid clinicians in planning the most appropriate therapeutic strategy. The differential diagnosis using power Doppler sonography is based on vascular characteristics. Adenomyosis is characterized by a preserved vascular texture supply that results in dilated spiral arteries running perpendicular toward the myometrium into the endometrial surface. Leiomyomata exhibits a vascular tree that typically circumscribes the solid mass. 2D transvaginal power Doppler angiography should be used to improve diagnostic sensitivity and facilitate appropriate therapeutic intervention.

The levonorgestrel-releasing intrauterine system (IUS), Mirena, has been approved in Europe for contraception since 1990. Because of the suppressive effect of levonorgestrel on the endometrium, Mirena has also been proven to be effective for the management of menorrhagia and dysmenorrhea, and as a progestin component in postmenopausal hormone therapy. It was introduced in Taiwan in 1995 as an alternative therapy for idiopathic menorrhagia. Many cases of menorrhagia are caused by adenomyosis, and Mirena was, therefore, introduced for the treatment of adenomyosis in Taiwan.

The current study is designed to evaluate the best treatment modality for treatment of adenomyosis clinical by assessment of dysmenorrhea and or chronic pelvic pain by visual analogue scale and menstrual blood loss by menstrual diary, imaging by ultrasound and Doppler indices.

ELIGIBILITY:
Inclusion Criteria:

1. Women have dysmenorrhoea and/or chronic pelvic pain secondary to adenomyosis.
2. Planning for birth spacing for at least 2 years.
3. Patient aged between 20-45 years old.
4. Ultrasonographic and Doppler examination suggestive of adenomyosis.
5. Living in a nearby area to make follow-up reasonably possible.

Exclusion Criteria:

1. Pregnancy
2. Evidence of defective coagulation.
3. History or evidence of malignancy.
4. Hyperplasia in the endometrial biopsy.
5. Incidental adnexal abnormality on ultrasound.
6. Contraindications to COCs.
7. Absolute contraindication of LNG-IUS insertion.
8. Previous endometrial ablation or resection
9. Uninvestigated postcoital bleeding
10. Untreated abnormal cervical cytology

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Visual analogue score (VAS) for dysmenorrhea or chronic pelvic pain will be measure before after use LNG_IUS and COCs. | 6 month

SECONDARY OUTCOMES:
Menstrual blood loss: assessment of blood loss, measured at the beginning of intervention and for 3 months | 6 month